CLINICAL TRIAL: NCT00598000
Title: Quality of Life and Pain Outcomes Following Video-Assisted Thoracic Surgery (VATS) Anatomic Lung Resection Versus Thoracotomy and Anatomic Lung Resection
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 05-006
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Lung Cancer; Quality of Life; Video-assisted Thoracic Surgery (VATS); Thoracotomy
Keywords: Lung cancer; Quality of Life; VATS; thoracotomy; 05-006
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Determine the impact, in terms of quality of life (QOL), of minimally invasive, video-assisted thoracic surgery (VATS)
  Interventions: Behavioral: questionnaires
- 2: Determine the impact, in terms of quality of life (QOL), in traditional thoracotomy and anatomic lung resection in early stage lung cancer.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — QOL Measures- The following measures will be administered at Pre-Op, First Post-Op Visit 4, 8, 12 months Post-Op.
  Brief Pain Inventory and daily analgesic log- enrollment, patients will fill out the BPI preoperatively, postoperative days 2 to 4, initial, 4-month, 8-month and 12-month postoperative visits.
  Groups: 1
Behavioral: questionnaires — QOL Measures- The following measures will be administered at Pre-Op, First Post-Op Visit 4, 8, 12 months Post-Op.
  Brief Pain Inventory and daily analgesic log- enrollment, patients will fill out the BPI preoperatively, postoperative days 2 to 4, initial, 4-month, 8-month and 12-month postoperative visits.
  Groups: 2

SUMMARY:
The purpose of this study is to see if different types of surgery for lung cancer have different effects on quality of life and pain. What we learn from this study may help us find new ways to improve the quality of life of lung cancer patients who have surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed or suspected clinical stage I non small cell lung cancer (including carcinoid tumors) based on standard staging (CT, PET, ± mediastinoscopy).
* Patients offered a VATS anatomic lung resection or a standard, posterolateral thoracotomy and anatomic lung resection at MSKCC.
* Patients cannot have had prior therapy, including surgery for the current lesion, systemic chemotherapy or external beam radiotherapy.
* KPS ≥ 70.
* Synchronous primaries within one lobe.

Exclusion Criteria:

* Patients who have already undergone the planned operation.
* Patients who cannot tolerate segmentectomy or lobectomy.
* Patients with locally advanced or metastatic disease found either preoperatively or at the time of operation.
* Patients who are non- English speaking
* Patients with multi-focal disease
* Patients with con-current cancers
* Patients with benign disease.
* Patients who are unwilling or unable to return to Memorial Sloan-Kettering Cancer Center for postoperative follow-up for the first year following their operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MSKCC Clinics
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2005-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Determine the postoperative change in QOL and level of pain in patients with clinical stage I NSCLC undergoing VATS anatomic lung resection and for patients with clinical stage I NSCLC undergoing thoracotomy and anatomic lung resection | conclusion of study

SECONDARY OUTCOMES:
Compare early postoperative analgesic requirements between the VATS and thoracotomy groups. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Rizk, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org